CLINICAL TRIAL: NCT01962948
Title: A Phase I/II Trial of Weekly Paclitaxel In Combination With Ganetespib In Patients With Recurrent, Platinum-Resistant Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Paclitaxel and Ganetespib in Treating Patients With Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study drug is no longer supplied by grantor.
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GYN-064; NCI-2013-01416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB#13-028/ERP-GYN-064 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2022-06-24 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Taxes; STA 9090

STUDY DESIGN:
Intervention Model Description: Phase I Treatment: Paclitaxel IV given over 1 hour at 80 mg/m2 days 1, 8 and 15 of a 28-day cycle. PLUS ganetespib IV at a starting dose of 100 mg/m2 on days 1, 8 and 15 of a 28-day cycle. Ganetespib escalation will follow a modified 3+3 design and escalate from 100mg/m2 to 125mg/m2 to 150mg/m2. Phase II Treatment: Paclitaxel IV given over 1 hour at 80 mg/m2 days 1, 8 and 15 of a 28-day cycle. PLUS ganetespib IV at MTD/MED from Phase I on days 1, 8 and 15 of a 28-day cycle.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1: 100 mg/m2 ganetespib, 80 mg/m2 paclitaxel (Experimental): Patients receive paclitaxel IV over 1 hour and ganetespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Ganetespib escalation will follow a modified 3+3 design and escalate from 100mg/m2 to 125mg/m2 to 150mg/m2.
  Interventions: Drug: paclitaxel; Drug: ganetespib; Other: laboratory biomarker analysis
- Phase I: 125 mg/m2 ganetespib, 80 mg/m2 paclitaxel (Experimental): Patients receive paclitaxel IV over 1 hour and ganetespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Ganetespib escalation will follow a modified 3+3 design and escalate from 100mg/m2 to 125mg/m2 to 150mg/m2.
  Interventions: Drug: paclitaxel; Drug: ganetespib; Other: laboratory biomarker analysis
- Phase I: 150 mg/m2 ganetespib, 80 mg/m2 paclitaxel (Experimental): Patients receive paclitaxel IV over 1 hour and ganetespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Ganetespib escalation will follow a modified 3+3 design and escalate from 100mg/m2 to 125mg/m2 to 150mg/m2.
  Interventions: Drug: paclitaxel; Drug: ganetespib; Other: laboratory biomarker analysis
- Phase II: MTD/MED of ganetespib, 80 mg/m2 paclitaxel (Experimental): Paclitaxel IV given over 1 hour at 80 mg/m2 days 1, 8 and 15 of a 28-day cycle. PLUS ganetespib IV at MTD/MED from Phase I on days 1, 8 and 15 of a 28-day cycle.
  Interventions: Drug: paclitaxel; Drug: ganetespib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: ganetespib — Given IV
  Other Names: Hsp90 inhibitor STA-9090; STA-9090
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of ganetespib when given together with paclitaxel and to see how well they work in treating patients with recurrent ovarian, fallopian tube, or primary peritoneal cancer. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Ganetespib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving paclitaxel and ganetespib may be an effective treatment for ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the recommended Phase II dose of ganetespib with weekly paclitaxel. (Phase I) II. Probability of surviving progression-free for at least 6 months after initiating therapy. (Phase II) III. Clinical response rate (partial and complete responses as defined by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria). (Phase II)

SECONDARY OBJECTIVES:

I. Determine the nature and degree of toxicity of ganetespib and weekly paclitaxel in this cohort of patients as measured by the frequency and severity of adverse reactions. (Phase I) II. Determine the nature and degree of toxicity of ganetespib and weekly paclitaxel in this cohort of patients as measured by the frequency and severity of adverse reactions encountered. (Phase II) III. Duration of progression-free survival. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of ganetespib followed by a phase II study.

Patients receive paclitaxel intravenously (IV) over 1 hour and ganetespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed recurrent epithelial ovarian, fallopian tube or primary peritoneal cancers who have received up to two prior treatment regimens
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria version (v.) 1.1
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation, or extended therapy administered after completion of initial chemotherapy; patients must be considered platinum resistant or refractory according to standard Gynecologic Oncology Group (GOG) criteria, i.e., have had a treatment-free interval following platinum of less than 12 months, have persistent disease at the completion of primary platinum-based therapy or have progressed during platinum-based therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< normal institutional limits
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) (serum glutamic oxaloacetic transaminase [SGOT]/serum glutamate pyruvate transaminase [SGPT]) =< 2 times institutional normal limits
* Creatinine =< normal institutional limits OR
* Creatinine clearance >= 60 Ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ability and willingness to comply with scheduled visits, treatment plan, laboratory assessments and other study procedures
* Ability to understand and willingness to sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent document

Exclusion Criteria:

* Patients who have had surgery, chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have toxicity that has not recovered to =< grade 1 from adverse events due to agents administered more than 4 weeks earlier (with the exception of alopecia); patients may not be receiving any other investigational agents
* Histologic diagnosis of a benign or borderline tumor ('tumor of low malignant potential') or of a malignant tumor of non-epithelial origin (such as a germ cell tumor, sex-cord stromal tumor) of the ovary, fallopian tube or peritoneum
* Patients with known brain metastases
* History of allergic reactions to Cremophor EL, paclitaxel or its components
* Prior history of >= grade 2 neurotoxicity or any other toxicity requiring discontinuation of taxane therapy that has not resolved to =< grade 1, with the exception of alopecia
* Diagnosis of another malignancy within two years before the first dose, or previously treated for another malignancy with evidence of residual disease, with the exception of a synchronous endometrial cancer; carcinoma in situ will not be considered as malignancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, known serious cardiac illness or psychiatric illness/social situations that would limit compliance with study requirements; known serious cardiac illness or medical conditions include, but are not limited to:

  * History of documented congestive heart failure (CHF), New York Heart Association (NYHA) class II/III/IV, with a history of dyspnea, orthopnea, or edema that requires current treatment with angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, beta blockers, or diuretics

    * NOTE: use of these medications for the treatment of hypertension is allowed
  * Screening QTc (QT interval corrected for heart rate) > 470 msec or history of QT (cardiac interval from start of Q wave to end of T wave) prolongation while taking other medications
  * High-risk uncontrolled arrhythmias (ventricular arrhythmias, high-grade atrioventricular [AV]-block, supra-ventricular arrhythmias that are not adequately rate-controlled)
  * Arrhythmias that require current treatment with the following anti-arrhythmic drugs: flecainide, moricizine, or propafenone
  * Current coronary artery disease with a history of myocardial infarction, angioplasty, or coronary bypass surgery within the preceding 6 months, or angina pectoris that has been symptomatic within the preceding 6 months
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Martina-Smaldone, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: 125 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel; Phase 1: 150 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel: Patients receive paclitaxel IV over 1 hour and ganetespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Ganetespib escalation will follow a modified 3+3 design and escalate from 100mg/m2 to 125mg/m2 to 150mg/m2.
Period: Overall Study
Arm/Group | Phase 1: 100 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase 1: 125 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase 1: 150 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase II: MTD/MED of Ganetespib, 80 mg/m2 Paclitaxel
Started | 3 | 3 | 6 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 0
Not completed — Study was closed because grantor stopped supplying study drug. Study did not progress to Phase II. | 3 | 3 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Study was closed because grantor stopped supplying study drug. Study did not progress to Phase II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: 100 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase 1: 125 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase 1: 150 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase II: MTD/MED of Ganetespib, 80 mg/m2 Paclitaxel | Total
Number analyzed (Participants) | 3 | 3 | 6 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4 | 0 | 8
  >=65 years | 1 | 1 | 2 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 0 | 12
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 2 | 3 | 6 | 0 | 11
  Black or African American | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose of Ganetespib With Weekly Paclitaxel, Based on the Incidence of Dose-limiting Toxicity (DLT) Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 (Phase I)
Time Frame: Up to 28 days
Measure: Number; unit: mg/m2 ganetespib
Groups:
- Treatment (Paclitaxel, Ganetespib): Patients receive paclitaxel IV over 1 hour and ganetespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  paclitaxel: Given IV
  ganetespib: Given IV
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Paclitaxel, Ganetespib)
Number analyzed (Participants) | 12
mg/m2 ganetespib | 150

2. Primary Outcome: Progression-free Survival at 6 Months (Phase II)
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed at 6 months
Population: The study was suspended prematurely due to halt in drug production and data were not analyzed
Arm/Group | Treatment (Paclitaxel, Ganetespib)
Number analyzed (Participants) | 0

3. Primary Outcome: Response Rate Defined as the Proportion of Patients With a Best Response of Complete Response (CR) or Partial Response (PR) Per RECIST v. 1.1 (Phase II)
Time Frame: Up to 4 years
Population: The study was suspended prematurely due to halt in drug production and data were not analyzed
Arm/Group | Treatment (Paclitaxel, Ganetespib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Progression-free Survival (Phase II)
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 4 years
Population: The study was suspended prematurely due to halt in drug production and data were not analyzed
Arm/Group | Treatment (Paclitaxel, Ganetespib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2.5 years
Description: Study was closed because grantor stopped supplying study drug. Study did not progress to Phase II.
Arm/Group | Phase 1: 100 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase 1: 125 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase 1: 150 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel | Phase II: MTD/MED of Ganetespib, 80 mg/m2 Paclitaxel
All-Cause Mortality (participants affected / at risk) | 3/3 | 1/3 | 4/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 100 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel (N=3) | Phase 1: 125 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel (N=3) | Phase 1: 150 mg/m2 Ganetespib, 80 mg/m2 Paclitaxel (N=6) | Phase II: MTD/MED of Ganetespib, 80 mg/m2 Paclitaxel (N=0)
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 4 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascite (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 5 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 3 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Hypertension (Cardiac disorders) | 2 | 0 | 3 | 0
Type II Diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gerd (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hearing loss (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 — PE right lung
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0
Hot flashes (General disorders) | 1 | 0 | 0 | 0
Edema (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 — limbs
Depression (Psychiatric disorders) | 1 | 0 | 2 | 0
Neck pain (General disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Brittle finger nails (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Oral thrush (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ecchymosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — IV site at forearm
Jitters (General disorders) | 0 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0
Sweats (General disorders) | 0 | 0 | 2 | 0
Heart palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Bleeding
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Back pain (General disorders) | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscle aches (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rib pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Shakiness (General disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT01962948/Prot_SAP_001.pdf